CLINICAL TRIAL: NCT01473446
Title: Traditional Versus Goal Directed Perioperative Fluid Therapy in High Risk Patients. A Randomized, Assessor-blinded Study
Brief Title: Traditional Versus Goal Directed Perioperative Fluid Therapy in High Risk Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High exclusion rate
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/947/REK Vest
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2013-03

CONDITIONS: Postoperative Complications
Keywords: Goal directed fluid therapy; perioperative fluid therapy; LiDCOrapid; Postoperative outcome; Open abdominal surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard monitoring. Initial optimization of fluid status is performed by pulse, BP and anaesthesiologist assessment with Ringer acetate. Followed by an infusion of 10ml/kg/t Ringer acetate. Urinary output and blood pressure is used as a surrogate parameter: the infusion rate is increased by a fall in blood pressure or urine output <0.5ml/kg/t. Bleeding replaced with HES 1:1, otherwise see table for fluid therapy page 9. Vasoactive agents (noradrenaline / phenylephrine) is given if the anesthesiologist considers this necessary. Postoperative give 1000ml Glucose 5%. HES or Ringer when low blood pressure, eventually noradrenaline as vasoactive agent.
- Goal directed fluid therapy (Experimental)
  Interventions: Procedure: Goal directed fluid therapy guided by LiDCOrapid

INTERVENTIONS:
Procedure: Goal directed fluid therapy guided by LiDCOrapid — Standard monitoring. The patient is connected to the LiDCOrapid monitor via an arterial line placed in a.radialis. A bolus of 500 ml Ringer acetate is given before anesthesia. If the stroke volume (SV) increases more than 10%, repeat the procedure until the SV is not increasing. After that, induction of anesthesia.
  Maintenance fluid is given as Ringer acetate 2ml/kg/t. Continuous monitoring of stroke volume variation (SVV). If SVV> 10%, give a fluid bolus 6ml/kg Ringer acetate. Repeat until SVV <10%. Bleeding is being replaced 1:1 with hydroxyethyl starch. SAG by bleeding >1000ml. By fall in blood pressure and SVV <10%, start vasoactive treatment with epinephrine. Postoperative is given Glucose 5% 80ml/h.
  Arms: Goal directed fluid therapy

SUMMARY:
Is goal directed fluid therapy reducing postoperative complications in comparison to traditional fluid therapy for gastro surgical ASA III/IV patients?

The investigators compare two groups of patients: one group receives goal directed fluid therapy guided by LiDCOrapid stroke volume variation (SVV), the other gets the "traditional" fluids, ie the current regime.

ELIGIBILITY:
Inclusion Criteria:

* Adult ASA class III & IV (high risk) patients
* >18 years
* scheduled for gastrointestinal surgery involving laparotomy
* Both elective and emergency cases

Exclusion Criteria:

* Atrial fibrillation
* Mental impairment, unable to give informed consent
* Severe aortic or mitral stenosis
* Type of surgery: Liver surgery, transthoracic oesophagectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 5 days after surgery

SECONDARY OUTCOMES:
Length of hospital stay | 3 month after surgery
Complications until discharge and readmission within 30 days | 3 month after surgery
Mortality within 30 days and 3-month after surgery | 3 month after surgery
Renal function | 5 days after surgery
  defined by RIFLE criteria
Vasoactive agents need | 3 month after surgery
  Difference in the number of patients in need of vasoactive agents, during surgery and in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Ib Jammer, MD, Study Chair — Helse Bergen HF, Norway
Locations (3):
- Oulu University Hospital, Department of Anesthesia and Intensive Care, Oulu, Finland
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger Universityhospital, Division for medical service, anesthesia and intensive care, Stavanger

REFERENCES:
- [Derived] Jammer I, Tuovila M, Ulvik A. Stroke volume variation to guide fluid therapy: is it suitable for high-risk surgical patients? A terminated randomized controlled trial. Perioper Med (Lond). 2015 Jul 22;4:6. doi: 10.1186/s13741-015-0016-x. eCollection 2015. PMID 26203353